CLINICAL TRIAL: NCT04619901
Title: How Parents (and Their Child if They Continue Their Life) Fare After a Decision of Palliative Care Has Been Taken in the Neonatal Period
Brief Title: Palliative Care in Maternity and Neonatology
Acronym: VESPAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_14; 2018-A01226-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-10-14; First posted 2020-11-06 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Neonatal Critical Care
Keywords: Palliative care; Maternity; newborn; parents
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents only
  Interventions: Other: Semi-structured interviews; Other: Questionnaire; Other: following Scales
- Children and Parents
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Semi-structured interviews — Exploring the psychological and social impact on parents of a palliative care decision concerning their child in the neonatal period
  Groups: Parents only
Other: Questionnaire — Assessing the neuro-developmental evolution of children and understanding the determinants of the psychological and social impact of palliative care decisions on parents
Other: following Scales — Scales : Hospital Anxiety and Depression, Intolerance to Uncertainty, and Brief COPE.
  Groups: Parents only

SUMMARY:
Palliative care is now an accepted principle in most maternity and neonatology wards, however not much is known about its psychological and social consequences on families. Some children continue their life after a palliative care decision has been taken. In France, quality of life and the neuro-developmental evolution of newborns who continue their life after a palliative care decision has been taken, have never been studied.

ELIGIBILITY:
Inclusion Criteria:

* Father and/or Mother of a child, who is alive or not, for whom a decision of palliative care has been made in the neonatal period
* Under the care of one of the Level 3 Maternity Centers in the North and Pas-de-Calais departments (Arras, Lens, Lille, Valenciennes) since 2018
* Written consent of the two legal guardians of the child allowing the collection of data concerning the child
* Written consent of the parent(s) participating to this study by completing the parental questionnaires

Exclusion Criteria:

* Medico-legal complaint underway
* Parents who do not understand French
* Parents or children who are under legal protection (guardianship, curatorship)
* Parents or children who are not Social Security beneficiaries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children and parents followed in pediatric unit whom a decision of palliative care has been made in the neonatal period
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Semi Structured interview | 24 months after palliative care decision
  Parents : Exploring the psychological and social impact of the palliative care decision 2 hours semi structured interviews will be done to describe the psychological and social impact a decision of palliative care concerning their newborn infant has on parents.

SECONDARY OUTCOMES:
Ages and Stages Questionnaire (ASQ) - Clinical Examination of Child | 24 months after palliative care decision
  Child : Neuro-Developmental Assessment
Semi Structured Interview | 24 months after palliative care decision
  Parents : Determinants of the psychological and social impact of the palliative care decision
Hospital Anxiety and Depression Scale (HADS) | 24 months after palliative care decision
  Parents :Psychometric Measure of Anxiety and Depression The scale allows to detect anxiety and depression using 14 items rated from 0-3.
Intolerance to Uncertainty Scale (EEI) | 24 months after palliative care decision
  Parents : Psychometric Measure of Intolerance to Uncertainty This questionnaire contains 27 items measuring emotions, cognitions and behaviours in ambiguous situations, the consequences of being uncertain and attempts to control the future.Items are rated on a Likert scale from 1 ("Not at all matching") to 5 ("Very matching"). The total share is obtained by adding the items.
Brief COPE | 24 months after palliative care decision
  Parents : Psychometric Measure of Coping Strategies The Brief-COPE is a 28 item self-report questionnaire withs scoring and interpretation: Positive reframing / Planning/ Humor / Religion/Self-blame

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Storme, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - CH ARRAS, Arras
  - CH LENS, Lens
  - Hop Jeanne de Flandre Chu Lille, Lille
  - CH Valenciennes, Valenciennes